CLINICAL TRIAL: NCT01439945
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Magnesium Supplements to Reduce Menopausal Hot Flashes
Brief Title: Magnesium Oxide in Treating Postmenopausal Women With Hot Flashes and a History of Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N10C2; NCCTG-N10C2; CDR0000711021 (Registry Identifier: PDQ (Physician Data Query)); NCI-2011-03537 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2011-09-22; First posted 2011-09-23 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer; Cancer Survivor; Hot Flashes
Keywords: hot flashes; cancer survivor; breast cancer
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes | interventions — Magnesium Oxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I (Experimental): Patients receive a low-dose of magnesium oxide orally (PO) daily (QD).
  Interventions: Drug: magnesium oxide
- Arm II (Experimental): Patients receive a high-dose of magnesium oxide PO QD.
  Interventions: Drug: magnesium oxide
- Arm III (Placebo Comparator): Patients receive a low-dose of placebo PO QD.
  Interventions: Other: placebo
- Arm IV (Placebo Comparator): Patients receive a high-dose of placebo PO QD.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: magnesium oxide — Given PO
  Arms: Arm I; Arm II
Other: placebo — Given PO
  Arms: Arm III; Arm IV

SUMMARY:
RATIONALE: Magnesium oxide may help relieve hot flashes symptoms in women with a history of breast cancer.

PURPOSE: This randomized clinical trial studies how well a high-dose or a low-dose of magnesium oxide works compared to placebo in treating menopausal women with hot flashes and a history of breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the efficacy of magnesium oxide on hot flashes in women with a history of breast cancer.

Secondary

* Evaluate the side-effect profile of magnesium oxide in this study population.
* Evaluate the effect of magnesium oxide on the secondary outcomes hot flash frequencies, hot flash severities, toxicities (including diarrhea), and hot flash-related daily interference on activities.
* Evaluate the effect of magnesium oxide on the change of magnesium level (for the first 150 patients).

OUTLINE: This is a multicenter study. Patients are stratified according to age (18-49 years vs ≥ 50 years), current tamoxifen and/or selective estrogen receptor modulator (yes vs no), current aromatase inhibitor (yes vs no), and daily frequency of hot flashes (4-9 vs ≥ 10). Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive a low-dose of magnesium oxide orally (PO) daily (QD).
* Arm II: Patients receive a high-dose of magnesium oxide PO QD.
* Arm III: Patients receive a low-dose of placebo PO QD.
* Arm IV: Patients receive a high-dose of placebo PO QD. In all arms, treatment continues for 8 weeks in the absence of unacceptable toxicity.

Some patients may continue or crossover to receive magnesium for 4 more weeks.

Patients complete the Hot Flash Diary daily for 9 weeks beginning 1 week before treatment. They also complete the Symptom Experience Questionnaire, the Profile of Mood States (POMS), and Hot Flash-Related Daily Interference Scale (HFRDIS) questionnaires periodically during study treatment.

Patients undergo blood sample collection at baseline and at the end of weeks 5 and 9 for serum magnesium level analysis.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Women with a history of breast cancer (currently without malignant disease)
* Bothersome hot flashes (defined by their occurrence ≥ 28 times per week and of sufficient severity to make the patient desire therapeutic intervention)
* Presence of hot flashes for ≥ 30 days prior to study registration
* Willingness to provide the biologic specimens as required by the protocol
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Women who are postmenopausal as defined by absence of a period in the past 12 months or bilateral oophorectomy

  * Women with at least one ovary but without a uterus should be deemed postmenopausal by either age over 55 or a combination of estrogen within a postmenopausal range (per local lab) and FSH over 40 mIU/mL
  * No women of childbearing potential or who are premenopausal
* Creatinine clearance > 30 mL/min
* Ability to complete questionnaire(s) by themselves or with assistance
* ECOG performance status 0 or 1
* No history of allergic or other adverse reaction to magnesium
* No diabetes
* No patients with conditions that are implicated in decreased absorption of magnesium (e.g., Crohn disease, ETOH abuse)
* No patients who have diarrhea where magnesium might make it worse (per provider discretion)

PRIOR CONCURRENT THERAPY:

* None of the following current (≤ 28 days prior to registration) or planned therapies (tamoxifen, raloxifene, or aromatase inhibitors are allowed, but the patient must have been on a constant dose for ≥ 28 days and must not be expected to stop the medication during the study period):

  * Antineoplastic chemotherapy (trastuzumab or lapatinib are allowed)
  * Androgens
  * Estrogens (any delivery route)
  * Progestational agents
* No prior use of magnesium for hot flashes
* No current or planned use of gabapentin (for any reasons) or antidepressants (for any reasons) or other agents for treating hot flashes (except stable dose of vitamin E is allowed as long as it was started > 30 days prior to study registration and are to be continued through the study period; soy is allowed, if it is planned to be continued at the same dose during the study period)
* No current use of magnesium for any indication (except one standard multiple vitamin dose is allowed per day)
* Not taking diuretics, corticosteroids, bile acid sequestrants, and other prescription and over-the-counter medications that may affect magnesium levels
* No current (≤ 7 days prior to registration) or planned use of other non-drug therapies for managing hot flashes, such as acupuncture or yoga (use of these therapies for other reasons is allowed)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2011-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Loprinzi, MD, Principal Investigator — Mayo Clinic
Locations (283):
- United States (283):
  - Fairbanks Cancer Treatment Center at Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Herbert D. Kerman Regional Oncology Center - Daytona Beach, Daytona Beach, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Kauai Medical Clinic, Lihue, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Oncare Hawaii, Incorporated - Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - St. Francis Hospital Cancer Care Services, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Cancer Center - West Lakes, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Central Care Cancer Center at Carrie J. Babb Cancer Center, Bolivar, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Goldschmidt Cancer Center, Jefferson City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Lovelace Medical Center - Downtown, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Park Ridge Hospital, Hendersonville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Mount Carmel Hospital East, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Southern Ohio Medical Center Cancer Center, Portsmouth, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson AFB, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - Carolina Blood and Cancer Care Associates, PA, Lancaster, South Carolina
  - Carolina Blood and Cancer Care, Rock Hill, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Pacific Medical Center, Seattle, Washington
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After the double blind phase patient were allowed to re-registered on the Optional Continuation Phase of the study. This phase lasted up to 4 weeks of treatment following either 800 or 1200 mg/day treatment group.
Groups:
- Low Dose Magnesium Oxide (800 mg/Day): Week 2:
  Patients take one 400 mg tablet of magnesium oxide orally (PO) daily (QD).
  Week 3:
  Patients take two 400 mg tablet of magnesium oxide orally (PO) daily (QD).
  Weeks 4-9:
  Patients take two 400 mg tablet of magnesium oxide orally (PO) daily (QD).
- High Dose Magnesium Oxide (1200 mg/Day): Week 2:
  Patients take one 400 mg tablet of magnesium oxide orally (PO) daily (QD).
  Week 3:
  Patients take two 400 mg tablet of magnesium oxide orally (PO) daily (QD).
  Weeks 4-9:
  Patients take three 400 mg tablet of magnesium oxide orally (PO) daily (QD).
- Low Dose Placebo: Week 2:
  Patients take one placebo tablets orally (PO) daily (QD).
  Week 3:
  Patients take two placebo tablets daily (QD).
  Weeks 4-9:
  Patients take two placebo tablets daily (QD).
- High Dose Placebo: Week 2:
  Patients take one placebo tablets orally (PO) daily (QD).
  Week 3:
  Patients take two placebo tablets daily (QD).
  Weeks 4-9:
  Patients take three placebo tablets daily (QD).
Period: Double-Blind Treatment Phase
Arm/Group | Low Dose Magnesium Oxide (800 mg/Day) | High Dose Magnesium Oxide (1200 mg/Day) | Low Dose Placebo | High Dose Placebo
Started | 97 | 96 | 48 | 48
Completed | 93 | 91 | 45 | 46
Not Completed | 4 | 5 | 3 | 2
Not completed — Withdrawal by Subject | 3 | 3 | 3 | 1
Not completed — Ineligible | 1 | 2 | 0 | 1
Period: Optional Continuation Phase
Arm/Group | Low Dose Magnesium Oxide (800 mg/Day) | High Dose Magnesium Oxide (1200 mg/Day) | Low Dose Placebo | High Dose Placebo
Started | 72 | 44 | 0 | 0
Completed | 72 | 44 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Patients registered to the High Dose Placebo and Low Dose Placebo are combined for treatment analysis.
  Week 2:
  Patients take one placebo tablets orally (PO) daily (QD).
  Week 3:
  Patients take two placebo tablets daily (QD).
  Weeks 4-9:
  Patients take two or three placebo tablets daily (QD).
- Total: Total of all reporting groups
Arm/Group | Low Dose Magnesium Oxide (800 mg/Day) | High Dose Magnesium Oxide (1200 mg/Day) | Placebo | Total
Number analyzed (Participants) | 93 | 91 | 91 | 275
Age, Customized [Count of Participants; unit: Participants]
  Age Group: 18-49 years | 15 | 15 | 15 | 45
  Age Group: >=50 | 78 | 76 | 76 | 230
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 91 | 91 | 275
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 93 | 91 | 91 | 275

OUTCOME MEASURES:

1. Primary Outcome: The Intra-patient Changes of Weekly Hot Flash Activity From Baseline During the Treatment Period.
Description: The primary endpoint is the intra-patient changes of weekly hot flash activity from baseline during the treatment period. The hot flash activity will be measured by the weekly average hot flash score, which is a composite entity of both frequency and severity of hot flashes.
  The hot flash severity is graded from 1 to 4 (1=mild, 2=moderate, 3=severe, and 4=very severe). The daily hot flash score is computed by multiplying the mean grade of severity by the frequency during every 24 hour period. Therefore, a score of zero is the lowest possible score and can be interpreted as having no hot flashes. The weekly hot flash score was calculated by adding all scores for the week.
  The mean Hot Flash Score for each week for each group is reported and a repeated measures analysis is reported comparing each dose level group to the Placebo group.
Time Frame: Baseline to Week 8
Population: All patients that began protocol treatment and completed the Hot Flash Diary were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Dose Magnesium Oxide (800 mg/Day) | High Dose Magnesium Oxide (1200 mg/Day) | Placebo
Number analyzed (Participants) | 88 | 88 | 91
units on a scale
  Baseline: number analyzed (Participants) | 81 | 81 | 83
  Baseline | 16.02 (9.62) | 15.35 (10.53) | 17.28 (10.84)
  Week 1: number analyzed (Participants) | 81 | 78 | 86
  Week 1 | 14.28 (9.26) | 14.47 (11.10) | 15.52 (10.51)
  Week 2: number analyzed (Participants) | 79 | 78 | 85
  Week 2 | 12.68 (8.87) | 12.59 (10.01) | 13.29 (9.46)
  Week 3: number analyzed (Participants) | 78 | 76 | 83
  Week 3 | 12.29 (9.79) | 11.32 (10.72) | 12.34 (9.98)
  Week 4: number analyzed (Participants) | 78 | 73 | 82
  Week 4 | 11.73 (10.35) | 10.14 (8.61) | 12.02 (9.57)
  Week 5: number analyzed (Participants) | 75 | 67 | 79
  Week 5 | 11.77 (10.86) | 9.73 (9.19) | 11.63 (9.61)
  Week 6: number analyzed (Participants) | 71 | 67 | 79
  Week 6 | 11.61 (10.46) | 9.44 (8.99) | 11.17 (8.78)
  Week 7: number analyzed (Participants) | 71 | 67 | 78
  Week 7 | 11.92 (11.26) | 9.37 (9.24) | 10.71 (8.68)
  Week 8: number analyzed (Participants) | 69 | 66 | 79
  Week 8 | 12.17 (10.88) | 9.06 (8.87) | 11.42 (10.32)
Statistical Analysis 1: Comparison: Low Dose Magnesium Oxide (800 mg/Day) vs Placebo; Test type: Superiority or Other; p = 0.13, ANOVA; Weekly hot flash score was treated as a repeated measure for each patient
Statistical Analysis 2: Comparison: High Dose Magnesium Oxide (1200 mg/Day) vs Placebo; Test type: Superiority or Other; p = 0.67, ANOVA; Weekly hot flash score was treated as a repeated measure for each patient

2. Secondary Outcome: Weekly Frequency of Hot Flashes as Measured by the Hot Flash Diary During the Treatment Period
Description: As part of the Hot Flash Diary, the number of hot flashes was recorded for each patient for each week. For this endpoint, the mean number of hot flashes for each group is reported. A repeated measure analysis comparing each dose level group and the Placebo is reported.
Time Frame: Baseline to Week 8
Population: All patients that began protocol treatment and completed the Hot Flash Diary were included in this analysis.
Measure: Mean (Standard Deviation); unit: number of hot flashes
Arm/Group | Low Dose Magnesium Oxide (800 mg/Day) | High Dose Magnesium Oxide (1200 mg/Day) | Placebo
Number analyzed (Participants) | 88 | 88 | 91
number of hot flashes
  Baseline: number analyzed (Participants) | 81 | 81 | 83
  Baseline | 8.48 (4.34) | 7.55 (3.89) | 8.89 (4.52)
  Week 1: number analyzed (Participants) | 81 | 78 | 86
  Week 1 | 7.83 (4.34) | 7.15 (4.13) | 8.04 (4.59)
  Week 2: number analyzed (Participants) | 79 | 78 | 85
  Week 2 | 7.12 (4.18) | 6.51 (4.19) | 7.26 (4.65)
  Week 3: number analyzed (Participants) | 78 | 76 | 83
  Week 3 | 6.73 (4.41) | 5.87 (4.21) | 6.97 (4.82)
  Week 4: number analyzed (Participants) | 78 | 73 | 82
  Week 4 | 6.39 (4.51) | 5.34 (3.76) | 6.73 (4.44)
  Week 5: number analyzed (Participants) | 75 | 67 | 79
  Week 5 | 6.31 (4.70) | 5.15 (4.00) | 6.45 (4.33)
  Week 6: number analyzed (Participants) | 71 | 67 | 79
  Week 6 | 6.34 (4.56) | 4.95 (4.04) | 6.37 (4.30)
  Week 7: number analyzed (Participants) | 71 | 67 | 78
  Week 7 | 6.43 (4.68) | 4.92 (4.13) | 6.18 (4.23)
  Week 8: number analyzed (Participants) | 69 | 66 | 79
  Week 8 | 6.61 (4.58) | 4.88 (4.02) | 6.38 (4.67)
Statistical Analysis 1: Comparison: Low Dose Magnesium Oxide (800 mg/Day) vs Placebo; Test type: Superiority or Other; p = 0.25, ANOVA; Weekly number of hot flashes were treated as a repeated measure for each patient
Statistical Analysis 2: Comparison: High Dose Magnesium Oxide (1200 mg/Day) vs Placebo; Test type: Superiority or Other; p = 0.55, ANOVA — Weekly number of hot flashes were treated as a repeated measure for each patient

3. Secondary Outcome: Frequency and Maximum Grade of Adverse Events Reported Via the CTCAE 4.0 During the Treatment Period.
Description: Frequency and severity of adverse events reported by patients in weekly Symptom Experience Questionnaire and evaluated through clinical assessment by NCI CTCAE v3.0. The number of patients reporting grade 3 or higher events are reported in this outcome measure. For a full list of all events, please refer to the Adverse Events section of this report.
Time Frame: Baseline to Week 8
Population: All patients that started protocol treatment and were evaluated for adverse events are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Magnesium Oxide (800 mg/Day) | High Dose Magnesium Oxide (1200 mg/Day) | Placebo
Number analyzed (Participants) | 92 | 93 | 92
Participants
  Grade 3+ Adverse Event | 5 | 1 | 2
  Grade 4+ Adverse Event | 0 | 0 | 0

4. Secondary Outcome: The Change of Severity of Symptoms as Measured the Symptom Experience Questionnaire From Baseline to Treatment Termination
Description: We will use the Symptom Experience Questionnaire (SEQ) to evaluate the specific impact of the study treatment on the effect hot flashes have on various life activities such as work, social, leisure and relationships. The questionnaire is 14 questions and is based on a 0="Not at all" to 10="As bad as it can be" scale. The change of severity of symptoms as measured by the SEQ from baseline to treatment termination will be first summarized by descriptive statistics as a percent change from baseline.
Time Frame: Baseline to week 8
Population: All patients that started treatment and completed the Symptom Experience Questionnaire at baseline and Cycle 9 were included in this analysis.
Measure: Median (Full Range); unit: percentage change
Arm/Group | Low Dose Magnesium Oxide (800 mg/Day) | High Dose Magnesium Oxide (1200 mg/Day) | Placebo
Number analyzed (Participants) | 79 | 80 | 82
percentage change
  Stomach Pain | 0 [-40 to 60] | 0 [-30 to 30] | 0 [-60 to 40]
  Diarrhea | 0 [-50 to 20] | -5 [-90 to 50] | 0 [-80 to 50]
  Nausea | 0 [-50 to 70] | 0 [-70 to 50] | 0 [-60 to 50]
  Dizziness | 0 [-20 to 50] | 0 [-80 to 50] | 0 [-30 to 20]
  Decreased Appetite | 0 [-10 to 50] | 0 [-20 to 20] | 0 [-40 to 30]
  Fatigue | 0 [-100 to 70] | 0 [-40 to 70] | 0 [-30 to 80]
  Muscle Weakness | 0 [-80 to 50] | 0 [-50 to 70] | 0 [-60 to 30]
  Abnormal Sweating | 10 [-80 to 90] | 10 [-50 to 80] | 10 [-80 to 80]
  Constipation | 0 [-70 to 70] | 0 [-50 to 100] | 0 [-50 to 70]
  Muscle/Joint Aches | 5 [-90 to 80] | 10 [-80 to 60] | 0 [-30 to 50]
  Trouble Sleeping | 10 [-40 to 80] | 40 [-50 to 70] | 10 [-40 to 100]
  Negative mood change | 0 [-50 to 50] | 0 [-30 to 60] | 0 [-70 to 80]
  Trouble Concentrating | 0 [-50 to 60] | 0 [-30 to 50] | 0 [-40 to 70]
  Distress | 10 [-60 to 100] | 20 [-60 to 70] | 10 [-60 to 80]

5. Secondary Outcome: The Change of Daily Interference as Measured by the Hot Flash Related Daily Interference Scale (HFRDIS) From Baseline to Treatment Termination.
Description: We will use the Hot Flash Related Daily Interference Scale (HFRDIS) (SEQ) to evaluate the specific effect of hot flashes have on various life activities such as work, social, leisure and relationships while receiving treatment. The questionnaire is 10 questions and is based on a 0="Do not interfere" to 10="Completely interfere" scale. The weekly score is the summation of these 10 questions and therefore ranges from 0 to 100. The total change in severity of symptoms is calculated by subtracting the week 8 score from the baseline. Therefore, values below zero indicate a worsening of symptoms and values above zero indicate an improvement and has a maximum range of -100 to 100. A gatekeeper procedure, following a fixed-sequence hypothesis testing method, was used to examine the higher dose of magnesium vs. placebo first and then the lower dose of magnesium vs. placebo, if the former was statistically significant.
Time Frame: Baseline to week 8
Population: All patients that began treatment and completed the HFRDI questionnaire at baseline and week 8 were used in this analysis.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | High Dose Magnesium Oxide (1200 mg/Day) | Placebo
Number analyzed (Participants) | 73 | 74
units on a scale | 7 [-26 to 45] | 8.5 [-41 to 74]
Statistical Analysis 1: Comparison: High Dose Magnesium Oxide (1200 mg/Day) vs Placebo; Test type: Superiority or Other; p = 1.00, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: The Intra-patient Changes of Magnesium Level From Baseline to the End of Treatment Period Between Magnesium Oxide and Placebo Arms.
Description: The intra-patient changes of magnesium level from baseline to the end of treatment period between magnesium oxide and placebo arms will be compared using a repeated measures model.
  Serum magnesium concentrations will be performed prior to study medication usage and during the last week of blinded study use. These will be obtained in the first 150 patients. Mean change in serum magnesium concentrations will be compared between the 3 study arms to determine whether there are any apparent changes in the patients receiving placebos vs the two magnesium doses.
Time Frame: Baseline to week 8
Population: All patients that started protocol treatment and had serum magnesium levels obtained at baseline and week 9 were included in this analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Low Dose Magnesium Oxide (800 mg/Day) | High Dose Magnesium Oxide (1200 mg/Day) | Placebo
Number analyzed (Participants) | 69 | 74 | 72
mg/dL | 0.0 (0.2) | 0.1 (0.2) | 0.0 (0.2)
Statistical Analysis 1: Comparison: Low Dose Magnesium Oxide (800 mg/Day) vs Placebo; Test type: Superiority or Other; p = 0.47, Kruskal-Wallis
Statistical Analysis 2: Comparison: High Dose Magnesium Oxide (1200 mg/Day) vs Placebo; Test type: Superiority or Other; p = 0.09, Kruskal-Wallis

ADVERSE EVENTS:
Description: All patients that began treatment and were assessed for adverse events (AEs) are reported. In the Low Dose arm, 97 patients were randomized, 5 were never assessed for AEs. In the High Dose arm, 96 patients were randomized, 3 patients were never assessed for AEs. In the placebo arms, 96 patients were randomized, 4 were never assessed for AEs. This leaves 92, 93, and 92 patients on Low Dose, High Dose and Placebo arms respectively assessed for Adverse events.
Groups:
- Optional Continuation Phase: After the double blind phase patient questionnaire booklet has been completed and returned to the investigator, the patient will be told whether she was on magnesium or placebo. If the patient wishes to continue or start the magnesium, and healthcare provider approves that this is an appropriate option, she may be registered on the Optional Continuation Phase of the study. This phase will last up to 4 weeks of treatment following either 800 or 1200 mg/day treatment group.
Arm/Group | Low Dose Magnesium Oxide (800 mg/Day) | High Dose Magnesium Oxide (1200 mg/Day) | Placebo | Optional Continuation Phase
Serious Adverse Events (participants affected / at risk) | 0/92 | 1/93 | 0/92 | 0/116
Other Adverse Events (participants affected / at risk) | 67/92 | 40/93 | 31/92 | 40/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Magnesium Oxide (800 mg/Day) (N=92) | High Dose Magnesium Oxide (1200 mg/Day) (N=93) | Placebo (N=92) | Optional Continuation Phase (N=116)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Magnesium Oxide (800 mg/Day) (N=92) | High Dose Magnesium Oxide (1200 mg/Day) (N=93) | Placebo (N=92) | Optional Continuation Phase (N=116)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (5) | 0 (0) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (7) | 2 (3) | 3 (3) | 1 (2)
Bloating (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (13) | 1 (1) | 1 (2) | 1 (4)
Diarrhea (Gastrointestinal disorders) | 52 (137) | 26 (66) | 21 (37) | 32 (52)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (5) | 2 (5) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (5) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 10 (21) | 6 (7) | 3 (4) | 4 (7)
Oral pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (11) | 1 (1) | 3 (5) | 2 (5)
Autoimmune disorder (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (8) | 1 (1) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (10) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (14) | 1 (1) | 0 (0) | 2 (5)
Headache (Nervous system disorders) | 4 (6) | 2 (2) | 3 (3) | 1 (2)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (7) | 3 (4) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Dysmenorrhea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 2 (2) | 1 (1) | 2 (8) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less